CLINICAL TRIAL: NCT00208091
Title: An Open Label Evaluation of MIDI to Quantify Performance Change in Subjects With Musician's Dystonia After Treatment With Botulinum Toxin Type B (Myobloc ®).
Brief Title: Quantifying Musical Performance After Treatment With Myobloc in Musician's Dystonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Solstice Neurosciences (Industry)
Responsible Party: Principal Investigator, Seth Pullman, Professor of Clinical, Department of Neurology, Movement Disorders, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB2808
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Focal Dystonia
Keywords: Myloboc; Botulinum Toxin Type B; Focal Dystonia; Musicians; Muscle Relaxants; Motor Impairments; Motor Performance; Tremor; Abnormal Postures
MeSH Terms: conditions — Dystonic Disorders; Muscle Hypotonia; Tremor | interventions — rimabotulinumtoxinB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botulinum toxin, type B (Experimental): Diluted botulinum toxin (500 Units/0.1 ml) is injected to the affected muscle(s) through a hollow core needle using electromyographic guidance. Dosage according to muscle(s) and symptom severity. Injection occurs at first visit only, after neurological evaluation.
  Interventions: Drug: Botulinum toxin, type B

INTERVENTIONS:
Drug: Botulinum toxin, type B — Diluted botulinum toxin (500 Units/0.1 ml) is injected to the affected muscle(s) through a hollow core needle using electromyographic guidance. Dosage according to muscle(s) and symptom severity. Injection occurs at first visit only, after neurological evaluation.
  Other Names: Myobloc

SUMMARY:
This study uses a computerized method of musical instrument digital interface (MIDI) quantification of performance before and after treatment with botulinum toxin type B (Myobloc ®, Solstice Neurosciences). Myobloc is a purified and diluted form of botulinum toxin used medically to relax unwanted muscle spasms and movements. The aim of the study is to determine the feasibility of quantifying change in performance following treatment.

DETAILED DESCRIPTION:
Dystonia represents a group of clinical disorders characterized by various combinations of sustained involuntary muscle contractions, abnormal postures and movements, tremors and pain. Dystonia can occur at rest but is more likely to appear during voluntary activity.

Focal dystonia affects one body area and includes blepharospasm, oromandibular dystonia, spasmodic dysphonia, torticollis, and limb dystonia. Focal dystonia typically presents as task-specific muscle spasms or "occupational cramps" in which learned or repetitive motor tasks (such as writing or playing a musical instrument) trigger muscle spasms and interfere with performance while other actions remain normal. Writer's cramp is the most common form of idiopathic limb dystonia [1-3] where involuntary muscle activity and abnormal postures affect the arms and hands, but virtually any part of the body may be affected, even the lips when playing a woodwind or brass instrument [4]. Patients may develop two focal dystonias but rarely does focal dystonia progress to more generalized forms.

As originally defined by Oppenheim [5], dystonia refers to the slow, sustained, writhing, contorting movements of dystonia musculorum deformans. Dystonic movements, however, are often rapid [6] and this can be a cause for misdiagnosis. Electromyography (EMG) may be helpful in corroborating dystonia, but is not essential for diagnostic purposes. Nerve conduction studies, short and long loop reflexes and analysis of motor units are normal [7, 8]. Ballistic movements, which are normally tri-phasic in pattern with alternating agonist-antagonist bursts, may show disrupted patterns with co-contraction of agonist and antagonist muscles and excessively long EMG bursts in dystonia [3].

Dystonic spasms are intriguing in that they may be suppressed (or triggered) by sensory input such as postural change, tactile stimuli, alternative movements or even thought processes [9]. Studies are revealing that the involuntary muscle spasms may be due, at least in part, to abnormal sensory processing of spindle afferent information [10-12]. This may help explain the nature of these sensory "tricks" as well as why the effect of treatment using botulinum toxin usually outlasts the weakness it creates.

Though the pathophysiology of musicians' dystonia has yet to be determined fully, the motor learning associated with playing a musical instrument probably results in both functional and structural changes in the brain [13]. This plastic reorganization, including the rapid unmasking of existing neural circuitry and the establishment of new connections, is probably fundamental to the accomplishment of skillful playing, but also may result in focal, task-specific dystonia. When musicians get dystonia, their playing abilities can become severely compromised, to the point where they may not be able to perform professionally, and possibly not even teach. While botulinum toxin injections can be highly successful in allowing musicians to perform again, there are no objective methods to evaluate improvement.

Subtle dystonic abnormalities in motor control, therefore, particularly when they involve the arms, are difficult to ascertain with a high level of certainty. There are no truly objective measures of arm dystonia, and this is problematic because arm involvement can present so mildly as to go unnoticed by the examiner [14]. Furthermore, patients may not complain of mild finger or thumb cramping, arm twisting or shoulder elevation that could signify the presence of dystonia.

Clinical rating scales, even those that have been validated, do not detect subtle motor dysfunction or small changes after treatment [15] and certainly cannot determine improvement in musical performance. Metabolic imaging studies using positron emission tomography (PET) studies are emerging as helpful ancillary tests, but these are invasive and expensive. Furthermore, while PET studies have implicated that primary dystonia may be associated with relative hypermetabolism in the putamen [16], there have been conflicting reports [17]. Another major difficulty in the study of musician's dystonias has been lack of objective, quantifiable methods to assess degrees of dystonia severity or measure of treatment effects. Subjective and objective clinical rating scales with varying degrees of sophistication. Some subjective methods that have been used include subjective quantification usually using percentage improvement, also different various subjective rating scales using surveys.

This study tests a novel method devised for quantifying change in musical performance based on musical instrument digital interface (MIDI) data that will be able to directly rate or score changes in musical output. MIDI data include information on the note played, the time of onset, note duration, and note loudness. Note duration and loudness will be used in this study. It will be a quantitative, objective computerized evaluation that compares the patients' fine motor skills before and after treatment with Myobloc ®. It will be one of the first quantitative analyses of musical ability of its kind and could significantly impact the way musicians determine the efficacy of botulinum toxin treatment.

REFERENCES

1. Nutt JG, Muenter MD, Melton LJ, Aronson A, Kurland LT. Epidemiology of dystonia in Rochester, Minnesota. Adv Neurol 1988; 50: 361-5.
2. Sheehy MP, Marsden CD. Writers' cramp - a focal dystonia. Brain 1982; 105: 461-480.
3. Cohen LG, Hallett M. Hand cramps: clinical features and electromyographic patterns in a focal dystonia. Neurology 1988; 38: 1005-1012.
4. Frucht S, Fahn S, Ford B. French horn embouchure dystonia. Mov Disord 1999; 14: 171-3.
5. Oppenheim H. Uber eine eigenartige Krampfkrankheit des kindlichen und jungendichen Alters (dysbasia lordotica progressiva, dystonia musculorum deformans). Neurologie Centralblatt 1911; 30: 1090-1107.
6. Fahn S. Concept and classification of dystonia. In Fahn, S, Marsden, CD, Caln, DB, ed. Advances in Neurology: Dystonia 2. New York: Raven Press, 1988: 1-8.
7. Rothwell JC, Obeso JA, Day BL, Marsden CD. Pathophysiology of dystonias. In Desmedt, JE, ed. Advances in Neurology: Motor Control Mechanisms in Health and Disease. New York: Raven Press, 1983: 851-863.
8. Marsden CD, Rothwell JC. The physiology of idiopathic dystonia. Can J Neurol Sci 1987; 14: 521-527.
9. Greene PE, Bressman S. Exteroceptive and interoceptive stimuli in dystonia. Mov Disord 1998; 13: 549-51.
10. Tempel L, Perlmutter J. Abnormal vibration-induced cerebral blood flow responses in idiopathic dystonia. Brain 1990; 113: 691-707.
11. Kaji R, Rothwell JC, Katayama M, Tomoko I, Kubori T, Kohara N, Mezaki T, Shibasaki H, Kimura J. Tonic vibration reflex and muscle afferent block in writer's cramp. Ann Neurol 1995; 38: 155-162.
12. Koelman JHTM, Willemse RB, Bour LJ, Hilgevoord AAJ, Speelman JD, Ongerboer de Visser BW. Soleus H-reflex tests in dystonia. Mov Disord 1995; 10: 44-50.
13. Pascual-Leone A. The brain that plays music and is changed by it. Ann N Y Acad Sci 2001; 930: 315-29.
14. Bressman SB, de Leon D, Kramer PL, Ozelius LJ, Brin MF, Greene PE, Fahn S, Breakefield XO, Risch NJ. Dystonia in Ashkenazi Jews: Clinical characterization of a founder mutation. Ann Neurol 1994; 36: 771-777.
15. Burke RE, Fahn S, Marsden CD, Bressman SB, Moskowitz C, Friedman J. Validity and reliability of a rating scale for the primary torsion dystonias. Neurology 1985; 35: 73-77.
16. Eidelberg D, Moeller JR, Ishikawa T, Dhawan V, Spetsieris P, Przedborski S, Fahn S. The metabolic topography of idiopathic torsion dystonia. Brain 1995; 118: 1473-1484.
17. Karbe H, Holthoff VA, Rudolf J, Herholz K, Heiss WD. Positron emission tomography demonstrates frontal cortex and basal ganglia hypometabolism in dystonia. Neurology 1992; 42: 1540-1544.
18. Pullman SL. Limb dystonia: Use of botulinum toxin. In Jankovic, J, Hallett, M, ed. Therapeutic Use of Botulinum Toxin. New York: Marcel Dekker, 1994: 307-321.
19. Medical Research Council Aids to the Examination of the Peripheral Nervous System; Crown: London, 1976.
20. Pullman SL, Greene P, Fahn S, Pedersen SF. Approach to the treatment of limb disorders with botulinum toxin A. Experience with 187 patients. Arch Neurol 1996; 53: 617-24.
21. Cohen LG, Hallett M, Geller BD, Hochberg F. Treatment of focal dystonias of the hand with botulinum toxin injections. J Neurol Neurosurg Psychiatry 1989; 52: 355-363.
22. Trosch RM, Pullman SL. Botulinum toxin A injections for the treatment of hand tremors. Mov Disord 1994; 9: 601-9.

ELIGIBILITY:
Inclusion Criteria:

* Focal, task-specific dystonia clinically determined to be the result of a high level of musical skill and intensive performance history

Exclusion Criteria:

* Neurological disorders other than dystonia
* Patients who are clinically depressed, demented or otherwise unable to perform appropriately or sit through 1 hour of testing
* Patients who have undergone pallidotomy, thalamotomy or deep brain stimulator implantations
* Patients who have who recently have taken medications with extrapyramidal or tremorogenic side effects

Ages: 25 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Pullman, MD, Principal Investigator — Columbia University Medical Center, Department of Neurology
Locations (1):
- Neurological Institute, 710 W. 168th Street, NI-1112, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The dates of recruitment for this study were from April 2003 to May 2008. Both male and female subjects were included. Each subject must have been diagnosed with a focal, task-specific dystonia which was clinically determined to be the result of a high level of musical skill and intensive performance history to be included in the study.
Period: Overall Study
Arm/Group | Botulinum Toxin, Type B
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin, Type B
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.375 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Note Errors (Related to Errors in Duration)
Description: Note errors (related to errors in duration in msec) were obtained as measures of difference between the affected and unaffected hands--taking the musical instrument digital interface (MIDI) note output from four musical sequences of 8 to 16 notes played. It was calculated by averaging the sequences for each hand, and deriving the square root of the mean of the square of the differences (root mean square error, in msec) in MIDI.
Time Frame: Baseline and 6 weeks post-injection
Measure: Median (Standard Error); unit: msec
Groups:
- Note Errors (Related to Errors in Duration), Baseline: Note errors (related to errors in duration) were calculated as measures of difference between the affected and unaffected hand performing multiple scale sequences of 8 to 16 notes played. This was obtained by averaging sequences, note by note, for each hand and taking the square root of the mean of the square of the differences (root mean square error) in note duration.
- Note Errors (Related to Errors in Duration), Post-injection: Note errors 6 weeks after diluted botulinum toxin (500 Units/0.1 ml) was injected to the affected muscle(s) through a hollow core needle using electromyographic guidance. Dosages varied for each patient according to symptom severity and involved muscle(s).
Arm/Group | Note Errors (Related to Errors in Duration), Baseline | Note Errors (Related to Errors in Duration), Post-injection
Number analyzed (Participants) | 16 | 16
msec | 8.20 (8.49) | 5.79 (4.00)
Statistical Analysis 1: Comparison: Note Errors (Related to Errors in Duration), Baseline vs Note Errors (Related to Errors in Duration), Post-injection; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Note Errors (Related to Errors in Loudness)
Description: Note errors (related to errors in loudness) were obtained as a measure of difference between the affected and unaffected hands--taking the musical instrument digital interface (MIDI) note loudness data (decibels) from four musical sequences of 8 to 16 notes. It was calculated by averaging sequences for each hand and taking the square root of the mean of the square of the differences (root mean square error, in decibels) in MIDI notes.
Time Frame: Baseline and 6 weeks post-injection
Measure: Median (Standard Error); unit: decibels
Groups:
- Note Errors, Baseline: Note errors (related to errors in loudness) were calculated as a measure of difference between the affected and unaffected hand performing multiple scale sequences of 8 to 16 notes. This was obtained by averaging sequences, note by note, for each hand and taking the square root of the mean of the square of the differences (root mean square error) in note loudness.
- Note Errors, Post-injection: Note errors (related to errors in loudness) 6 weeks after diluted botulinum toxin (500 Units/0.1 ml) was injected to the affected muscle(s) through a hollow core needle using electromyographic guidance. Dosages varied for each patient according to symptom severity and involved muscle(s).
Arm/Group | Note Errors, Baseline | Note Errors, Post-injection
Number analyzed (Participants) | 16 | 16
decibels | 10.06 (1.28) | 8.43 (1.63)
Statistical Analysis 1: Comparison: Note Errors, Baseline vs Note Errors, Post-injection; Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Subjective Assessment Ratings of Change
Description: Each subject assessed his or her music playing performance change subjectively from -100 percent (fully worse) to 100 percent (fully better).
Time Frame: Baseline to 6 weeks after injection
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Post-injection Subjective Change: Subjective assessment 6 weeks after diluted botulinum toxin (500 Units/0.1 ml) was injected to the affected muscle(s) through a hollow core needle using electromyographic guidance. Dosages varied for each patient according to symptom severity and involved muscle(s).
Arm/Group | Post-injection Subjective Change
Number analyzed (Participants) | 16
percentage change | 30 (29.3)

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin, Type B
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No